CLINICAL TRIAL: NCT01245725
Title: A Randomized, Multicenter, Double-Blind, Study to Evaluate the Efficacy of Tirofiban HCl Versus Placebo in the Setting of Standard Therapies Among Subjects Undergoing Percutaneous Coronary Intervention
Brief Title: Aggrastat Truncated Length Against Standard Therapies in Percutaneous Coronary Intervention
Acronym: ATLAST-PCI
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was not initiated, change in clinical development
Sponsor: Medicure (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10002
Record Dates: First submitted 2010-11-12; First posted 2010-11-22 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Infarction; Acute Coronary Syndromes; Unstable Angina; Percutaneous Coronary Intervention
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Angina, Unstable | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tirofiban (Aggrastat) (Experimental)
  Interventions: Drug: Tirofiban (Aggrastat)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirofiban (Aggrastat) — Tirofiban (Aggrastat) will be dosed as a 25mcg/kg i.v. bolus followed by a 0.15mcg/kg/min i.v. infusion during a percutaneous coronary intervention plus two hours after the procedure.
  Patients will receive tirofiban (Aggrastat) on a background of oral anti-platelet agent(s) and either unfractionated heparin (50U/kg and repeat dosing guided per guidelines) or bivalirudin as per local practice and physician discretion.
  Arms: Tirofiban (Aggrastat)
Drug: Placebo — Placebo will be dosed as an i.v. bolus followed by an i.v. infusion during a percutaneous coronary intervention plus two hours after the procedure.
  Patients will receive placebo on a background of oral anti-platelet agent(s) and either unfractionated heparin (50U/kg and repeat dosing guided per guidelines) or bivalirudin as per local practice and physician discretion.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the efficacy of tirofiban (a 25mcg/kg i.v. bolus followed by a 0.15mcg/kg/min i.v. infusion during a percutaneous coronary intervention (PCI) plus two hours after the procedure) is more effective than placebo in the setting of standard therapies (e.g. aspirin, a thienopyridine, and unfractionated heparin or bivalirudin) among patients undergoing PCI, as assessed by the incidence of adverse cardiac ischemic events defined as death, myocardial infarction (MI), and urgent target vessel revascularization (uTVR) within 48 hours following study drug initiation.

A secondary objective of this study is to assess whether tirofiban (a 25mcg/kg i.v. bolus followed by a 0.15mcg/kg/min i.v. infusion during a PCI plus two hours after the procedure) is safe compared to placebo in the setting of standard therapies (e.g. aspirin, a thienopyridine, and unfractionated heparin or bivalirudin) among patients undergoing PCI, as assessed by the incidence of non-CABG-related TIMI major bleeding within 48 hours following study drug initiation.

Patient enrollment is pending.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age
2. Scheduled to undergo PCI with an approved device
3. Written informed consent

Exclusion Criteria:

1. Primary PCI for ST-elevation myocardial infarction (STEMI)
2. Prior PCI within 30 days
3. Prior GPIIb/IIIa use within 14 days
4. Prior enoxaparin use within 4 days
5. Prior STEMI within 30 days
6. In non-elective subjects, a rising troponin defined as a most recent pre-PCI sample greater than the sample immediately preceding it, as long as the two samples are separated by four or more hours and have been analyzed in the same hospital laboratory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
A composite incidence of death, myocardial infarction and urgent target vessel revascularization. | 48 hours

SECONDARY OUTCOMES:
The occurrence of myocardial infarction. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Steven V Manoukian, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Background] Topol EJ, Moliterno DJ, Herrmann HC, Powers ER, Grines CL, Cohen DJ, Cohen EA, Bertrand M, Neumann FJ, Stone GW, DiBattiste PM, Demopoulos L; TARGET Investigators. Do Tirofiban and ReoPro Give Similar Efficacy Trial. Comparison of two platelet glycoprotein IIb/IIIa inhibitors, tirofiban and abciximab, for the prevention of ischemic events with percutaneous coronary revascularization. N Engl J Med. 2001 Jun 21;344(25):1888-94. doi: 10.1056/NEJM200106213442502. PMID 11419425
- [Background] Valgimigli M, Percoco G, Barbieri D, Ferrari F, Guardigli G, Parrinello G, Soukhomovskaia O, Ferrari R. The additive value of tirofiban administered with the high-dose bolus in the prevention of ischemic complications during high-risk coronary angioplasty: the ADVANCE Trial. J Am Coll Cardiol. 2004 Jul 7;44(1):14-9. doi: 10.1016/j.jacc.2004.03.042. PMID 15234398
- [Background] Valgimigli M, Campo G, de Cesare N, Meliga E, Vranckx P, Furgieri A, Angiolillo DJ, Sabate M, Hamon M, Repetto A, Colangelo S, Brugaletta S, Parrinello G, Percoco G, Ferrari R; Tailoring Treatment With Tirofiban in Patients Showing Resistance to Aspirin and/or Resistance to Clopidogrel (3T/2R) Investigators. Intensifying platelet inhibition with tirofiban in poor responders to aspirin, clopidogrel, or both agents undergoing elective coronary intervention: results from the double-blind, prospective, randomized Tailoring Treatment with Tirofiban in Patients Showing Resistance to Aspirin and/or Resistance to Clopidogrel study. Circulation. 2009 Jun 30;119(25):3215-22. doi: 10.1161/CIRCULATIONAHA.108.833236. Epub 2009 Jun 15. PMID 19528337
- [Background] Valgimigli M, Campo G, Percoco G, Bolognese L, Vassanelli C, Colangelo S, de Cesare N, Rodriguez AE, Ferrario M, Moreno R, Piva T, Sheiban I, Pasquetto G, Prati F, Nazzaro MS, Parrinello G, Ferrari R; Multicentre Evaluation of Single High-Dose Bolus Tirofiban vs Abciximab With Sirolimus-Eluting Stent or Bare Metal Stent in Acute Myocardial Infarction Study (MULTISTRATEGY) Investigators. Comparison of angioplasty with infusion of tirofiban or abciximab and with implantation of sirolimus-eluting or uncoated stents for acute myocardial infarction: the MULTISTRATEGY randomized trial. JAMA. 2008 Apr 16;299(15):1788-99. doi: 10.1001/jama.299.15.joc80026. Epub 2008 Mar 30. PMID 18375998
- [Background] Valgimigli M, Tebaldi M. Safety evaluation of tirofiban. Expert Opin Drug Saf. 2010 Sep;9(5):801-19. doi: 10.1517/14740338.2010.507189. PMID 20670206
- [Background] Moliterno DJ; TENACITY Steering Committee and Investigators. A randomized two-by-two comparison of high-dose bolus tirofiban versus abciximab and unfractionated heparin versus bivalirudin during percutaneous coronary revascularization and stent placement: the tirofiban evaluation of novel dosing versus abciximab with clopidogrel and inhibition of thrombin (TENACITY) study trial. Catheter Cardiovasc Interv. 2011 Jun 1;77(7):1001-9. doi: 10.1002/ccd.22876. Epub 2011 Jan 11. PMID 21598351